CLINICAL TRIAL: NCT00636766
Title: Atherosclerotic Plaque Texture-Experimental and Clinical Study on the Diagnostic and Therapeutic Strategies of Atherosclerotic Plaque Vulnerability
Brief Title: Diagnosis and Therapy of Vulnerable Atherosclerotic Plaque
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Nikolaos Kadoglou, MD,PhD, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Factorial | Masking: None
Other Study IDs: 887/2005
Record Dates: First submitted 2008-03-11; First posted 2008-03-14 (Estimated); Last update posted 2012-11-02 (Estimated); Status verified 2012-11

CONDITIONS: Carotid Atherosclerosis; Stroke; Type 2 Diabetes; Metabolic Syndrome
Keywords: cardiovascular events
MeSH Terms: conditions — Carotid Artery Diseases; Stroke; Diabetes Mellitus, Type 2; Metabolic Syndrome | interventions — Atorvastatin; Rimonabant; Rosiglitazone; Metformin

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: atorvastatin; Drug: rimonabant; Drug: rosiglitazone; Drug: metformin

INTERVENTIONS:
Drug: atorvastatin — A:Experimental study of atherosclerosis B1:Effects of exercise on experimental atherosclerosis B2:Effects of exercise on high risk patients C1:Effects of statins on atherosclerotic plaque stability (experimental) C2:Effects of statins on atherosclerotic plaque stability (clinical) D:Effects of rosiglitazone and metformin on cardiovascular risk factors E:Effects of rimonabant on atherosclerotic plaque stability (experimental)
Drug: rimonabant — A:Experimental study of atherosclerosis B1:Effects of exercise on experimental atherosclerosis B2:Effects of exercise on high risk patients C1:Effects of statins on atherosclerotic plaque stability (experimental) C2:Effects of statins on atherosclerotic plaque stability (clinical) D:Effects of rosiglitazone and metformin on cardiovascular risk factors E:Effects of rimonabant on atherosclerotic plaque stability (experimental)
Drug: rosiglitazone — A:Experimental study of atherosclerosis B1:Effects of exercise on experimental atherosclerosis B2:Effects of exercise on high risk patients C1:Effects of statins on atherosclerotic plaque stability (experimental) C2:Effects of statins on atherosclerotic plaque stability (clinical) D:Effects of rosiglitazone and metformin on cardiovascular risk factors E:Effects of rimonabant on atherosclerotic plaque stability (experimental)
Drug: metformin — A:Experimental study of atherosclerosis B1:Effects of exercise on experimental atherosclerosis B2:Effects of exercise on high risk patients C1:Effects of statins on atherosclerotic plaque stability (experimental) C2:Effects of statins on atherosclerotic plaque stability (clinical) D:Effects of rosiglitazone and metformin on cardiovascular risk factors E:Effects of rimonabant on atherosclerotic plaque stability (experimental)

SUMMARY:
The aim of the present study is to examine the atherosclerotic plaque stability using in vivo and in vitro techniques and to investigate the influence of exercise, anti-diabetic, lipid-lowering and cannabinoids receptor antagonists on atherosclerotic plaque texture in patients with cardiovascular risk and animals prone to atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Carotid atherosclerosis
* Femoral atherosclerosis
* Cardiovascular risk

Exclusion Criteria:

* Heart failure
* Renal disease
* Liver disease
* Life-threatening diseases

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2005-09; Primary Completion 2007-12 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Ultrasound and immunohistochemical parameters of plaque stability; novel cardiovascular risk factors | 3 years

SECONDARY OUTCOMES:
Long-term cardiovascular outcomes | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Christos Liapis, Professor, Study Chair — University of Athens
Locations (1):
- General Hospital of Thessaloniki "Hippokratio", Thessaloniki, Greece

REFERENCES:
- [Derived] Kadoglou NP, Moulakakis KG, Papadakis I, Ikonomidis I, Alepaki M, Spathis A, Karakitsos P, Lekakis J, Liapis CD. Differential effects of stent-graft fabrics on arterial stiffness in patients undergoing endovascular aneurysm repair. J Endovasc Ther. 2014 Dec;21(6):850-8. doi: 10.1583/14-4772MR.1. PMID 25453890
- [Derived] Moustardas P, Kadoglou NP, Katsimpoulas M, Kapelouzou A, Kostomitsopoulos N, Karayannacos PE, Kostakis A, Liapis CD. The complementary effects of atorvastatin and exercise treatment on the composition and stability of the atherosclerotic plaques in ApoE knockout mice. PLoS One. 2014 Sep 29;9(9):e108240. doi: 10.1371/journal.pone.0108240. eCollection 2014. PMID 25264981
- [Derived] Lambadiari V, Kadoglou NP, Stasinos V, Maratou E, Antoniadis A, Kolokathis F, Parissis J, Hatziagelaki E, Iliodromitis EK, Dimitriadis G. Serum levels of retinol-binding protein-4 are associated with the presence and severity of coronary artery disease. Cardiovasc Diabetol. 2014 Aug 21;13:121. doi: 10.1186/s12933-014-0121-z. PMID 25142320
- [Derived] Kadoglou NP, Tahmatzidis DK, Giannakoulas C, Kapelouzou A, Gkontopoulos A, Parissis J, Lampropoulos S, Kottas G. Serum levels of novel adipokines, omentin-1 and chemerin, in patients with acute myocardial infarction: KOZANI STUDY. J Cardiovasc Med (Hagerstown). 2015 May;16(5):341-6. doi: 10.2459/JCM.0000000000000053. PMID 25022935
- [Derived] Kadoglou NP, Lambadiari V, Gastounioti A, Gkekas C, Giannakopoulos TG, Koulia K, Maratou E, Alepaki M, Kakisis J, Karakitsos P, Nikita KS, Dimitriadis G, Liapis CD. The relationship of novel adipokines, RBP4 and omentin-1, with carotid atherosclerosis severity and vulnerability. Atherosclerosis. 2014 Aug;235(2):606-12. doi: 10.1016/j.atherosclerosis.2014.05.957. Epub 2014 Jun 8. PMID 24956535
- [Derived] Kadoglou NP, Fotiadis G, Lambadiari V, Maratou E, Dimitriadis G, Liapis CD. Serum levels of novel adipokines in patients with acute ischemic stroke: potential contribution to diagnosis and prognosis. Peptides. 2014 Jul;57:12-6. doi: 10.1016/j.peptides.2014.04.008. Epub 2014 Apr 24. PMID 24768795
- [Derived] Kadoglou NP, Sailer N, Fotiadis G, Kapelouzou A, Liapis CD. The impact of type 2 diabetes and atorvastatin treatment on serum levels of MMP-7 and MMP-8. Exp Clin Endocrinol Diabetes. 2014 Jan;122(1):44-9. doi: 10.1055/s-0033-1358762. Epub 2014 Jan 24. PMID 24464597